CLINICAL TRIAL: NCT04343053
Title: Patterns and Changes in Platelet Reactivity, Thrombotic Status and Endothelial Function in Hospitalized Patients with SARS-Cov-2 Infection
Brief Title: Pro-thrombotic Status in Patients with SARS-Cov-2 Infection
Acronym: ATTAC-Co
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Associate Professor, University Hospital of Ferrara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 250320
Record Dates: First submitted 2020-04-03; First posted 2020-04-13 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2

STUDY DESIGN:
Masking Description: Technicians performing assays will be blinded to stage of the infection and outcomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SARS-Cov-2 infection (Other): Single study group of patients with respiratory failure due to SARS-Cov-2 infection. Three blood samples will be collected at different stages of disease: early, defined as first 96 hours, mid, defined as time from 96 hours and 14 days, late. defined as >14 days
  Interventions: Other: SARS-Cov-2 infection

INTERVENTIONS:
Other: SARS-Cov-2 infection — blood sample withdrawal

SUMMARY:
The present study is ideated to prospectively investigate in patients with severe acute respiratory syndrome (SARS) due to Coronavirus 19 (SARS-Cov-2) infection and moderate-severe respiratory failure the patterns and changes in platelet reactivity, thrombotic status and endothelial function. The observed patterns and changes will be related with inflammatory status, myocardial injury and outcomes

DETAILED DESCRIPTION:
Preliminary evidences suggested that patients with SARS-Cov-2 infection and concomitant presence of cardiovascular risk factors (i.e. arterial hypertension) and/or cardiovascular history (i.e. prior myocardial infarction) are at poor prognosis. The first reports from China suggested in patients with SARS-Cov-2 infection a heightened inflammatory burden associated with significant changes in coagulative status (i.e. low platelet count, increased D-dimer) and dysfunction of micro-vessels in pulmonary circulation.

No data are available about patterns and changes in platelet reactivity, activation of coagulation factors and endothelial function during SARS-Cov-2 infection.

The present study is ideated to fill this gap. Patients with moderate to severe respiratory failure due to SARS-Cov-2 infection will be enrolled. One blood sample will be obtained from each patient at the early, mid and late stage of disease. Several markers of platelet, coagulation and endothelial function will be related with laboratory, clinical, electrocardiographic, imaging (transthoracic echocardiogram, pulmonary ultrasonography, computed tomography) and outcome data.

To better describe typical patterns of disease regarding inflammation, platelet function and coagulation alteration, data from cases will be compared with control groups negative for SARS-CoV-2 infection, but with ST-segment elevation myocardial infarction or moderate-severe respiratory failure due to other agents.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate-severe respiratory failure (PaO2/FiO2 <200)
* Diagnosis of SARS-CoV-2 infection + one of the following

  1. invasive mechanical ventilation (cohort A)
  2. non invasive mechanical ventilation (cohort B)
  3. only oxygen support

Exclusion Criteria:

* Previous chronic use of P2Y12 inhibitors
* Need for chronic oral anti-coagulation therapy
* Know disorder of coagulation or platelet function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2023-11-12 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
on-treatment platelet reactivity | early stage of disease (first 96 hours)
  patterns and changes of platelet aggregation values assessed by light transmission aggregometry after arachidonic acid, adenosine diphosphate and thrombin receptor activating peptide stimuli
on-treatment platelet reactivity | mid stage of disease (96 hours - 14 days)
  patterns and changes of platelet aggregation values assessed by light transmission aggregometry after arachidonic acid, adenosine diphosphate and thrombin receptor activating peptide stimuli
on-treatment platelet reactivity | late stage of disease (>14 days)
  patterns and changes of platelet aggregation values assessed by light transmission aggregometry after arachidonic acid, adenosine diphosphate and thrombin receptor activating peptide stimuli

SECONDARY OUTCOMES:
apoptosis rate in human umbilical vein endothelial cells (HUVEC) | early stage of disease (first 96 hours)
  patterns and changes of the rate of apoptosis in HUVEC incubated with serum from patients enrolled in the study.
apoptosis rate in human umbilical vein endothelial cells (HUVEC) | mid stage of disease (96 hours - 14 days)
  patterns and changes of the rate of apoptosis in HUVEC incubated with serum from patients enrolled in the study.
Nitric oxide (NO) intracellular levels | late stage of disease (>14 days)
  patterns and changes of intracellular level of NO in HUVEC incubated with serum from patients enrolled in the study.
Nitric oxide (NO) intracellular levels | early stage of disease (first 96 hours)
  patterns and changes of intracellular level of NO in HUVEC incubated with serum from patients enrolled in the study.
Nitric oxide (NO) intracellular levels | mid stage of disease (96 hours - 14 days)
  patterns and changes of intracellular level of NO in HUVEC incubated with serum from patients enrolled in the study.
reactive oxygen species (ROS) levels | early stage of disease (first 96 hours)
  patterns and changes of ROS
reactive oxygen species (ROS) levels | mid stage of disease (96 hours - 14 days)
  patterns and changes of ROS
reactive oxygen species (ROS) levels | late stage of disease (>14 days)
  patterns and changes of ROS
coagulation factors levels | early stage of disease (first 96 hours)
  patterns and changes of the most important coagulation factors (i.e. tissue factor antigen pg/dL)
coagulation factors levels | mid stage of disease (96 hours - 14 days)
  patterns and changes of the most important coagulation factors (i.e. tissue factor antigen pg/dL)
coagulation factors levels | late stage of disease (>14 days)
  patterns and changes of the most important coagulation factors (i.e. tissue factor antigen pg/dL)
respiratory function | 6-month
  values of FEV1% as assessed by spirometry
respiratory function | 12-month
  values of FEV1% as assessed by spirometry
cardiac function | 6-month
  values of left ventricular ejection fraction as assessed by transthoracic echocardiogram
cardiac function | 12-month
  values of left ventricular ejection fraction as assessed by transthoracic echocardiogram
clinical outcome | 12-month
  occurrence of death, myocardial infarction, stroke and other major adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Savino Spadaro, MD, Principal Investigator — Intensive care unit; Gianluca Campo, MD, Principal Investigator — Cardiology Unit; Marco Contoli, MD, Principal Investigator — Pulmonology Unit
Locations (1):
- Azienda Ospedaliera Universitaria di Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Yes
After specific request to study PIs
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Scaramuzzo G, Ronzoni L, Campo G, Priani P, Arena C, La Rosa R, Turrini C, Volta CA, Papi A, Spadaro S, Contoli M. Long-term dyspnea, regional ventilation distribution and peripheral lung function in COVID-19 survivors: a 1 year follow up study. BMC Pulm Med. 2022 Nov 9;22(1):408. doi: 10.1186/s12890-022-02214-5. PMID 36352423
- [Derived] Contoli M, Papi A, Tomassetti L, Rizzo P, Vieceli Dalla Sega F, Fortini F, Torsani F, Morandi L, Ronzoni L, Zucchetti O, Pavasini R, Fogagnolo A, Volta CA, Bartlett NW, Johnston SL, Spadaro S, Campo G. Blood Interferon-alpha Levels and Severity, Outcomes, and Inflammatory Profiles in Hospitalized COVID-19 Patients. Front Immunol. 2021 Mar 9;12:648004. doi: 10.3389/fimmu.2021.648004. eCollection 2021. PMID 33767713
- [Derived] Spadaro S, Fogagnolo A, Campo G, Zucchetti O, Verri M, Ottaviani I, Tunstall T, Grasso S, Scaramuzzo V, Murgolo F, Marangoni E, Vieceli Dalla Sega F, Fortini F, Pavasini R, Rizzo P, Ferrari R, Papi A, Volta CA, Contoli M. Markers of endothelial and epithelial pulmonary injury in mechanically ventilated COVID-19 ICU patients. Crit Care. 2021 Feb 19;25(1):74. doi: 10.1186/s13054-021-03499-4. PMID 33608030
- [Derived] Campo G, Contoli M, Fogagnolo A, Vieceli Dalla Sega F, Zucchetti O, Ronzoni L, Verri M, Fortini F, Pavasini R, Morandi L, Biscaglia S, Di Ienno L, D'Aniello E, Manfrini M, Zoppellari R, Rizzo P, Ferrari R, Volta CA, Papi A, Spadaro S. Over time relationship between platelet reactivity, myocardial injury and mortality in patients with SARS-CoV-2-associated respiratory failure. Platelets. 2021 May 19;32(4):560-567. doi: 10.1080/09537104.2020.1852543. Epub 2020 Dec 3. PMID 33270471